CLINICAL TRIAL: NCT02070042
Title: Randomized Controlled Trial of Oxybutynin and Omega-3 Fatty Acid Supplementation Versus Oxybutynin and Placebo for Treatment of Overactive Bladder in Women
Brief Title: Oxybutynin and Omega-3 for OAB (Overactive Bladder)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participation
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13105-13-057
Record Dates: First submitted 2014-02-13; First posted 2014-02-24 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Oxybutynin; Omega -3 Fatty Acid
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Fatty Acids, Omega-3; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega- 3 Fatty Acid (Experimental): The patient will receive oxybutynin 5 mg twice daily (BID). The patients in the study group will receive a 0.9 gm capsule of Omega-3 BID. The amount of medication was chosen based on dosage used in prior studies and the current FDA recommendations to not exceed 2gm/day of omega-3 in dietary supplementation.
  Interventions: Drug: Omega 3 Fatty Acid
- Placebo (Placebo Comparator): Seagate® Extra Virgin Olive oil capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega 3 Fatty Acid — Trunature® Triple Strength Omega-3, given twice a day. Each capsule contains 647 mg Eicosapentaenoic Acid (EPA) and 253 mg Docosahexaenoic Acid (DHA).
  Arms: Omega- 3 Fatty Acid
Drug: Placebo — Placebo capsules (olive oil) twice a day
  Other Names: Olive Oil
  Arms: Placebo

SUMMARY:
We aim to evaluate whether the addition of Omega-3 fatty acids to oxybutynin, a standard first-line treatment for overactive bladder syndrome, will improve symptoms and quality of life. Secondarily, we will evaluate whether Omega-3 fatty acids help reduce the adverse effects of oxybutynin.

Hypothesis

* Primary: Omega-3 will enhance the beneficial role of oxybutynin in the treatment of overactive bladder (OAB)
* Secondary: Omega-3 will reduce the side effects of dry eyes and constipation associated with oxybutynin

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a troubling condition affecting over 17 million people in the U.S. with an estimated prevalence of 16.9% among women. The cost of this burden nationally was estimated at $66 billion in 2007. The morbidity of the disease impacts quality of life scores and increases risks of falls and fractures.

First-line therapeutic modalities for OAB focus on anticholinergic medications and behavioral modification. However, the indirect impact of these medications on the gut and salivary glands, have been troubling. Resultant side effect profiles with anticholinergic medications have caused a high rate of cessation, with some studies showing as low as 14% of patients still taking their medication at a one-year follow up. Given the burden and morbidity associated with this highly prevalent condition among women, our aim is to improve our therapeutic options, while possibly reducing subsequent side effects. As such, there is potential to revolutionize treatment for this condition.

Omega-3 fatty acids have been evaluated with success in treating many medical conditions. Specifically, diseases with an inflammatory component, such as Crohn's disease, ulcerative colitis, and rheumatoid arthritis have seen promising improvements with the addition of Omega-3 fatty acids. Other studies have shown a beneficial role in the treatment of dry eyes, depression, burn injuries, and even cancer. Although not previously explored in the setting of irritative bladder conditions, we believe that Omega-3 fatty acids may be helpful in interventions for OAB via several purported mechanisms.

Prostaglandin E2 (PGE2) and inflammation have both been implicated in the biochemistry of overactive bladder. Reduction in PGE2 may be paramount in reducing the symptoms of overactive bladder. In fact, a proposed mechanism of action of the success of anticholinergic medications, commonly first line treatment for OAB, is reduction of PGE2. Animal models have demonstrated that non-steroidal anti-inflammatory drugs (NSAIDs) can be used to decrease micturition frequency, which is thought to be a result of the anti-inflammatory process. In humans, anti-inflammatory medications have been shown to decrease nocturia and even cause urinary retention in high doses. Omega-3 fatty acids have been shown to have anti-inflammatory actions and the ability to reduce PGE2. We therefore, have reason to believe it may be an effective adjunct to current therapy to improve overactive bladder symptoms.

Additionally, Omega-3 fatty acids have been implemented in the treatment of dry eyes and animal studies have shown their role in increasing intestinal motility.Hence, we propose that Omega-3 fatty acids may help alleviate the common side effects of dry eyes and constipation associated with common anticholinergic therapies.

ELIGIBILITY:
Inclusion Criteria:

Women between the ages of 18-85; Desiring treatment for symptoms of urinary frequency, defined as >8 voids/day and/or nocturia > 1 void/night or urge incontinence episodes of >1/day

Exclusion Criteria:

Bleeding disorder; Uncontrolled diabetes; Hypotension; Liver disease, such as hepatitis A/B/C, cirrhosis, acute fatty liver, liver tumors; Post voiding residual (PVR) > 150 on more than one occasion; Uncontrolled narrow-angle glaucoma; Hematuria of unknown cause; Obstructive uropathy; Known hypersensitivity to study medications; Recent use of study/omega 3 or anticholinergic medication in the prior 3 weeks with an inability to discontinue this medication; Planning any surgery in the 6 weeks of study duration

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urinary voids per day | Baseline, 3 weeks and 6 weeks after enrollment
  The number of times the subjects urinates per day will be decreased

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Study Chair — TriHealth Inc.
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No